CLINICAL TRIAL: NCT07400718
Title: Head-to-Head Comparison Study Between Different FDA Registered Allergy Skin Test Applicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: QHSLab, Inc. (Industry)
Collaborators: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 33-098
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Allergy; Hypersensitivity, Immediate; Ig-E Mediated Food
Keywords: Allergy skin testing; Skin prick test; Multi-head skin test device; Device comparison; Diagnostic accuracy; Sensitivity and specificity; Intra-device variability
MeSH Terms: conditions — Hypersensitivity; Hypersensitivity, Immediate

STUDY DESIGN:
Intervention Model Description: This study employed a paired comparison design with each participant serving as their own control. Participants were assigned to one of two device comparison groups: (1) 10-head device comparison (AllerTest-10 vs. Skintestor OMNI, n=13), or (2) 8-head device comparison (AllerTest-8 vs. Multi-Test II, n=17). Within each comparison group, both devices were applied simultaneously-one to each forearm-with randomized left/right assignment. Each device was loaded with standardized histamine positive control and glycerin negative control. This within-subject design eliminates inter-subject variability in skin reactivity, providing robust paired comparisons of device performance on pain perception, control accuracy (sensitivity/specificity), and intra-device consistency.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- AllerTest Device (Experimental): Participants receive percutaneous allergy skin testing using an AllerTest multi-head device (either AllerTest-10 or AllerTest-8, manufactured by MedScience Research Group, Inc., distributed by ALK Abello, Inc.). The device is applied to one randomized forearm with a standardized histamine positive control (10 mg/mL histamine base) and a glycerin negative control (50% glycerin in saline). Outcomes measured include procedural pain (VAS 0-10), histamine wheal size at 15 minutes, glycerin wheal size at 15 minutes, sensitivity (proportion of histamine sites ≥3 mm), specificity (proportion of glycerin sites <3 mm), and intra-device variability (coefficient of variation across test heads).
  Interventions: Device: AllerTest-10 Multi-Head Skin Test Device; Device: AllerTest-8 Multi-Head Skin Test Device
- Comparator Device (Active Comparator): Participants receive percutaneous allergy skin testing using a comparator multi-head device (either Skintestor OMNI manufactured by Greer Laboratories, Inc., or Multi-Test II manufactured by Lincoln Diagnostics, Inc.). The device is applied simultaneously to the opposite forearm with identical standardized histamine positive control (10 mg/mL histamine base) and glycerin negative control (50% glycerin in saline). The same outcomes are measured to enable direct paired comparison: procedural pain (VAS 0-10), histamine wheal size at 15 minutes, glycerin wheal size at 15 minutes, sensitivity, specificity, and intra-device variability.
  Interventions: Device: Skintestor OMNI Multi-Head Skin Test Device; Device: Multi-Test II Multi-Head Skin Test Device

INTERVENTIONS:
Device: AllerTest-10 Multi-Head Skin Test Device — FDA-cleared 10-head percutaneous skin test applicator manufactured by MedScience Research Group, Inc., distributed by ALK Abello, Inc. The device consists of 10 individual test heads arranged in a linear array, each with a standardized needle length designed to penetrate the epidermis without drawing blood. Applied with standardized pressure for simultaneous delivery of 10 test substances (histamine and glycerin controls in this study). Single-use, disposable device.
  Other Names: AllerTest 10-head
  Arms: AllerTest Device
Device: Skintestor OMNI Multi-Head Skin Test Device — FDA-cleared 10-head percutaneous skin test applicator manufactured by Greer Laboratories, Inc. The device consists of 10 individual test heads arranged in a linear array for simultaneous application of multiple allergens and controls. Applied with standardized pressure for delivery of histamine and glycerin controls in this study. Single-use, disposable device.
  Arms: Comparator Device
Device: Multi-Test II Multi-Head Skin Test Device — FDA-cleared 8-head percutaneous skin test applicator manufactured by Lincoln Diagnostics, Inc. The device consists of 8 individual test heads arranged in a linear array for simultaneous application of multiple allergens and controls. Applied with standardized pressure for delivery of histamine and glycerin controls in this study. Single-use, disposable device.
  Arms: Comparator Device
Device: AllerTest-8 Multi-Head Skin Test Device — FDA-cleared 8-head percutaneous skin test applicator manufactured by MedScience Research Group, Inc., distributed by ALK Abello, Inc. The device consists of 8 individual test heads arranged in a linear array, each with a standardized needle length designed to penetrate the epidermis without drawing blood. Applied with standardized pressure for simultaneous delivery of 8 test substances (histamine and glycerin controls in this study). Single-use, disposable device.
  Arms: AllerTest Device

SUMMARY:
This clinical study, titled "Head-to-Head Comparison Study between Different FDA Registered Allergy Skin Test Applicators," aims to compare the reliability and clinical performance of three skin prick test (SPT) devices: Allertest™ Multiple Skin Test Applicator, Lincoln Multi-Test II, and Greer Skintestor OMNI Applicator. The primary objective is to evaluate the consistency and accuracy of these devices in allergy testing.

DETAILED DESCRIPTION:
Background and Rationale:

Percutaneous allergy skin testing remains the gold standard diagnostic method for IgE-mediated allergic disease. Multiple-head skin prick test (SPT) devices enable simultaneous application of multiple allergens, improving testing efficiency while potentially reducing patient discomfort. However, significant inter-device variability exists among commercially available devices, with important implications for diagnostic accuracy and clinical interpretation.

Intra-device variability-inconsistent responses across individual test heads within a single device-represents a particularly concerning phenomenon that may lead to physician misinterpretation and potentially inappropriate treatment decisions. Such variability can be attributed to manufacturing factors including tooling mold precision, molding equipment quality, and process controls during production. Prior research has demonstrated that devices with lower finished product variability exhibit improved clinical performance characterized by reduced false-positive reactions to negative controls.

Study Design:

This prospective, single-visit, head-to-head device comparison study employed a paired design in which each participant served as their own control, receiving testing with two devices simultaneously-one device applied to each forearm. This within-subject design minimizes inter-individual variability and provides robust comparative data.

Participants were allocated into two comparison groups based on device head configuration: a 10-head device comparison (n=13) and an 8-head device comparison (n=17). Device assignment to right versus left forearm was randomized. Testing personnel were blinded to solution contents (histamine versus glycerin) during application, and a separate evaluator blinded to device assignment recorded wheal measurements.

Study Procedures:

All testing was performed by trained personnel in accordance with standard percutaneous skin testing protocols. Histamine dihydrochloride (1 mg/mL; ALK-Abello) served as the positive control and glycerin solution (ALK-Abello) served as the negative control. Devices were applied to the volar forearm surfaces with standardized pressure and technique. Test sites were maintained at least 2 cm apart to prevent cross-contamination between histamine and glycerin reactions.

Wheal measurements were obtained 15-20 minutes post-application using the mean diameter method (average of longest diameter and its perpendicular midpoint), consistent with established international guidelines. Pain assessment was performed immediately following device application.

Statistical Considerations:

Paired comparisons between devices were analyzed using Wilcoxon signed-rank tests for continuous variables and McNemar's test for dichotomous outcomes. Intra-device variability was quantified using the coefficient of variation (CV) calculated across test heads, with lower values indicating greater consistency. Exact binomial (Clopper-Pearson) confidence intervals were calculated for sensitivity and specificity estimates. Statistical significance was set at α=0.05 (two-sided).

Clinical Significance:

This study addresses an important knowledge gap regarding comparative clinical performance of multi-head allergy testing devices. Results provide evidence-based data to inform device selection decisions that may impact diagnostic accuracy, patient comfort, and reliability of allergen identification in clinical allergy practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be entered into this study only if they meet all of the following criteria:

  1. Written and signed informed consent obtained before starting any protocol-specific procedures.
  2. Subjects willing to withhold antihistamines, Leukotriene antagonists and H2 antagonists for at least 1 week before testing to avoid masking the histamine reactions on the skin.
  3. Male or female between 18 to 60 65 years, inclusive.
  4. Ability to comply with the study procedures and visit schedule.

Exclusion Criteria:

* Patients will NOT be entered into this study if they meet any of the following criteria:

  1. Anaphylactic reaction (constitutional) after the previous skin test with the same allergen
  2. Acute fever
  3. Systemic disease with acute manifestation or decompensation
  4. Abnormal skin condition in the area to be tested (such as eczema sunburn condition after sunbathing)
  5. Pregnancy
  6. Presence of dermatographism, severe atopic dermatitis, or use of tricyclic antidepressants.
  7. Current use of beta-blockers
  8. Known hypersensitivity to any component of the test solutions (histamine or glycerin).
  9. Participation in another clinical study within 30 days before enrollment. Participation in another clinical study within 30 days before enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-11-12 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Pain Assessment Using Visual Analog Scale (VAS) | Immediately after device application (within 1 minute of skin test procedure)
  Procedural pain assessed immediately after device application using a 0-10 Visual Analog Scale (VAS), where 0 represents no pain and 10 represents unspeakable pain. Lower scores indicate less pain and better tolerability.
Sensitivity (Histamine Positive Control Performance) | 15 minutes after device application
  Proportion of histamine control sites producing wheal ≥3 mm diameter at 15 minutes post-application. A wheal of ≥3 mm is the standard threshold for a positive allergic reaction. Higher sensitivity indicates better device performance in reliably eliciting positive control responses. Calculated as: (number of histamine sites with wheal ≥3 mm) / (total number of histamine sites tested) × 100%.
Specificity (Glycerin Negative Control Performance) | 15 minutes after device application
  Proportion of glycerin control sites producing wheal <3 mm diameter at 15 minutes post-application. Glycerin should not produce a wheal response; a result <3 mm confirms appropriate negative control performance and absence of non-specific mechanical irritation. Higher specificity indicates better device performance. Calculated as: (number of glycerin sites with wheal <3 mm) / (total number of glycerin sites tested) × 100%.

SECONDARY OUTCOMES:
Intra-Device Variability | 15 minutes after device application
  Coefficient of variation (CV) of histamine wheal sizes across all test heads within each device, calculated as CV = (standard deviation / mean) × 100%. Lower CV values indicate greater consistency and precision across test heads within the same device. This measure reflects the reliability of allergen delivery across multiple heads of a single device application.
Mean Histamine Wheal Size | 15 minutes after device application
  Mean diameter (in millimeters) of wheals produced by histamine positive control across all test heads of each device. Wheal diameter measured using the mean diameter method (average of longest diameter and its perpendicular midpoint). Larger wheals indicate stronger positive control response.
Mean Glycerin Wheal Size | 15 minutes after device application
  Mean diameter (in millimeters) of wheals produced by glycerin negative control across all test heads of each device. Wheal diameter measured using the mean diameter method (average of longest diameter and its perpendicular midpoint). Smaller measurements (ideally 0 mm) indicate appropriate negative control performance with minimal non-specific irritation.
Proportion of Subjects with Clinically Significant Pain | Immediately after device application (within 1 minute of skin test procedure)
  Proportion of participants experiencing more than mild pain, defined as a score greater than 4 on the Visual Analog Scale (VAS) for pain. The VAS ranges from 0 (no pain) to 10 (unspeakable pain), with higher scores indicating worse pain. A threshold of >4 represents approximately 40% of the scale and indicates clinically meaningful discomfort. Lower percentages indicate better device tolerability across the study population. Reported as percentage with 95% exact binomial confidence intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- QHS Health center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Platts-Mills TA, Woodfolk JA. Rise in asthma cases. Science. 1997 Nov 7;278(5340):1001. doi: 10.1126/science.278.5340.997c. No abstract available. PMID 9381194
- [Result] Arbes SJ Jr, Gergen PJ, Elliott L, Zeldin DC. Prevalences of positive skin test responses to 10 common allergens in the US population: results from the third National Health and Nutrition Examination Survey. J Allergy Clin Immunol. 2005 Aug;116(2):377-83. doi: 10.1016/j.jaci.2005.05.017. PMID 16083793
- [Result] Cox L, Williams B, Sicherer S, Oppenheimer J, Sher L, Hamilton R, Golden D; American College of Allergy, Asthma and Immunology Test Task Force; American Academy of Allergy, Asthma and Immunology Specific IgE Test Task Force. Pearls and pitfalls of allergy diagnostic testing: report from the American College of Allergy, Asthma and Immunology/American Academy of Allergy, Asthma and Immunology Specific IgE Test Task Force. Ann Allergy Asthma Immunol. 2008 Dec;101(6):580-92. PMID 19119701
- [Result] Antunes J, Borrego L, Romeira A, Pinto P. Skin prick tests and allergy diagnosis. Allergol Immunopathol (Madr). 2009 May-Jun;37(3):155-64. doi: 10.1016/S0301-0546(09)71728-8. Epub 2009 Jul 23. PMID 19769849
- [Result] Bernstein IL, Li JT, Bernstein DI, Hamilton R, Spector SL, Tan R, Sicherer S, Golden DB, Khan DA, Nicklas RA, Portnoy JM, Blessing-Moore J, Cox L, Lang DM, Oppenheimer J, Randolph CC, Schuller DE, Tilles SA, Wallace DV, Levetin E, Weber R; American Academy of Allergy, Asthma and Immunology; American College of Allergy, Asthma and Immunology. Allergy diagnostic testing: an updated practice parameter. Ann Allergy Asthma Immunol. 2008 Mar;100(3 Suppl 3):S1-148. doi: 10.1016/s1081-1206(10)60305-5. No abstract available. PMID 18431959
- See also: Asthma and Allergy Foundation of America. CDC Fast Facts A-Z — https://aafa.org/asthma/asthma-facts/
- See also: Chronic Conditions: A Challenge for the 21st Century — http://www.partnershipforsolutions.org/DMS/files/chronic.pdf
- See also: United States Census Bureau — https://www.census.gov/quickfacts/fact/table/US/PST045224